CLINICAL TRIAL: NCT04516694
Title: Promoting Adolescent Investment In Diabetes Care
Acronym: InvesT1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Davene R. Wright, Faculty, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1540260
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes
Keywords: behavioral economics; financial incentive; diabetes; type 1 diabetes; adolescent; AYA; young adult
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Usual care reflects the standard treatment currently provided to T1D patients. All adolescent participants in the study will have access to the multidisciplinary care team including a diabetes provider, registered diabetes nurse, social worker, and nutritionist. Telephone consultations are available 24/7 as often as necessary between clinic visits.
- Gain-framed incentive (Experimental): Participants will start off with nothing at the beginning of the treatment period. For each day that participants' meet goals, value will be added to their incentive balance.
  All adolescent participants in the study will have access to the multidisciplinary care team including a diabetes provider, registered diabetes nurse, social worker, and nutritionist. Telephone consultations are available 24/7 as often as necessary between clinic visits.
  Interventions: Behavioral: Financial incentive (gain)
- Loss-framed incentive (Experimental): Participants will start off at the maximum incentive balance at the beginning of the treatment period and for each day that participants' fail to meet goals, value will be subtracted from their incentive balance over the 12-week.
  All adolescent participants in the study will have access to the multidisciplinary care team including a diabetes provider, registered diabetes nurse, social worker, and nutritionist. Telephone consultations are available 24/7 as often as necessary between clinic visits.
  Interventions: Behavioral: Financial incentive (loss)

INTERVENTIONS:
Behavioral: Financial incentive (gain) — Participants will receive a daily financial incentive framed as a gain with money allocated each day of adherence to a self-care coal. Participants will receive an additional weekly incentive for meeting a clinical outcome goal.
  Arms: Gain-framed incentive
Behavioral: Financial incentive (loss) — Participants will receive a daily financial incentive framed as a loss with money allocated up front and taken away each day of non-adherence to a self-care coal. An additional weekly incentive will be deducted for failure to meet a clinical outcome goal.
  Arms: Loss-framed incentive

SUMMARY:
Two financial incentive strategies targeting adolescents with type 1 diabetes will be compared to usual care for motivating adolescents to engage in improved self-care to manage their diabetes.

DETAILED DESCRIPTION:
Participants will be asked to choose a self-care goal relevant to the device(s) they use to manage their diabetes from a pre-defined list of self-care targets. A randomized 3 (treatment) x 3 (occasion) crossover design will be used to compare treatments that are administered to participants in a predetermined sequence. The intervention arms include financial incentives administered in a gain- and loss-frame for adherence to daily self-care goals. The control arm is usual care. Participants can also earn additional incentives for meeting clinical care goals such as an improvement in the percentage of time glucose levels are consistent with hyperglycemia (>180 mg/dL). The primary outcome will be HbA1c at 12 weeks compared to baseline. Secondary outcomes will include frequency of insulin administration, engagement in diabetes self-care (SCI-R), patient-reported outcomes (Problem Areas in Diabetes - Teen version and Diabetes Family Conflict Scale).

ELIGIBILITY:
Inclusion Criteria:

* >12 and ≤18 years old
* Diagnosed with type 1 diabetes ≥12 months
* Speaks English fluently
* Cognitively able to participate in incentive program and complete surveys.
* Have access to a mobile phone to receive goal-obtainment and incentive updates
* Receives diabetes-related clinical care from Seattle Children's Hospital Diabetes Clinic
* Have the ability to upload medical data remotely from home per usual care processes employed by Seattle Children's Hospital Diabetes Clinics

Exclusion Criteria:

* Patient is already participating in another research study to improve diabetes self-care and/or glycemic control
* Baseline daily average glucose checks are greater than 4 checks per day OR baseline daily CGM active wear is greater than 70% of the time AND baseline average insulin bolus score is greater than 3 times a day OR they do not use an insulin pump (or are unwilling to use a smart insulin pen)
* Patient refusal to participate (any age), or caregiver refusal to participate for patients less than 18 years of age
* Cognitively or physically unable to participate
* Patient is unable to speak in the English language
* Patient is unable to read in the English language
* Patient is a ward of the state
* Patient has severe comorbidities including other major chronic health conditions that significantly impact daily management demands or health outcomes

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-01-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 weeks
  Change in HbA1c from baseline to 12 weeks

SECONDARY OUTCOMES:
Glucose monitoring | 12 weeks
  Frequency of glucose monitoring
Insulin Administration | 12 weeks
  Insulin pumps and smart insulin pens track administration of all insulin manually delivered by the participant
SCI-R | 12 weeks
  The Self Care Inventory Revised is a 14-item self-report measure of perceived adherence to diabetes self-care recommendations
PAID-T | 12 weeks
  Problem Areas in Diabetes- Teen version
DFCS | 12 weeks
  Diabetes Family Conflict Scale
Time in Range | 12 weeks
  Evaluation of percentage of time spent in goal range via continuous glucose monitor system

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No